CLINICAL TRIAL: NCT01414868
Title: Could Leukotriene D4 Bronchial Provocation Test be a Clear Indicator for Predicting Therapeutic Outcomes of Leukotriene Receptor Antagonist A Pilot Study
Brief Title: Leukotriene D4 Bronchial Provocation Test (LTD4-BPT) as an Indicator for the Use of Leukotriene Receptor Antagonist (LTRA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Guangzhou Institute of Respiratory Disease, Guangzhou Institute of Respiratory Disease
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LTD4-BPT20110806
Record Dates: First submitted 2011-08-08; First posted 2011-08-11 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2009-12

CONDITIONS: Bronchial Asthma
Keywords: Leukotriene; leukotriene receptor antagonist; bronchial provocation test; therapeutic outcome
MeSH Terms: conditions — Asthma | interventions — Leukotriene Antagonists; montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: leukotriene receptor antagonist (montelukast) — montelukast (10 mg, once per night)
  Other Names: singulair

SUMMARY:
Background: Therapeutic outcomes of leukotriene receptor antagonist (LTRA) vary in asthmatics，and there's not an ideal and simple way for prediction at present.

Objective：To investigate whether leukotriene D4 bronchial provocation test (LTD4-BPT) could be an indicator of actual therapeutic outcome of LTRA.

Methods：A single centre, open-labeled trial was performed in 32 asthmatics with positive LTD4-BPT result for a month. All subjects were categorized according to airway responsiveness to leukotriene D4（PD20FEV1-LTD4）. Subjects received montelukast therapy (10mg, once per night), and reassessment was performed (3~5) days after withholding LTRA. The primary end-point was the difference in monthly PEFR. Secondary endpoints included the difference in FENO, PD20FEV1-LTD4, PD20FEV1-MCh, pre-test FEV1, ACT score, AQLQ symptom score, week 4 PEFmax and PEFmin as compared with week 1, gradual decrease in the use of salbutamol and the days without using salbutamol.

DETAILED DESCRIPTION:
Our primary goal was to determine whether LTD4-BPT could be a clear indicator for assessing efficacy of LTRA. Logistic regression model was adopted for statistical analysis. In this model, pre-treatment PD20FEV1-LTD4 represented anticipated efficacy. The median of PD20FEV1-LTD4 was used for classification of asthmatics, with a lower figure representing a better anticipated outcome. Various variables, including the difference in pre- and post- treatment FENO, PEFmax, PEFmin, PEFR, PD20FEV1 and asthma scores, were introduced in the model representing the actual efficacy of LTRA. We aimed to test whether there would be certain parameters that assist prediction of anticipated outcome.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged between 18 and 65，without acute upper respiratory tract infection for the past 2 weeks
* had a normal chest radiographic result
* had a baseline spirometry with the forced expiratory volume in one second (FEV1) of not less than 60% predicted
* had withheld leukotriene receptor antagonists (LTRA) for over 5 days
* oral glucocorticosteroid or anti-histamine for 3 days
* oral xanthenes or long-acting bronchodilators for 2 days
* inhaled corticosteroid or long-acting bronchodilator for a day as well as short-acting bronchodilator for 4 hours prior to the measurement

Exclusion Criteria:

* subjects had a fall of no less than 15% in FEV1 after repetitive forced respiration or a fall of no less than 20% in FEV1 after the inhalation of ethanol diluent control
* had a past confirmed history of respiratory disease other than bronchial asthma (COPD, bronchiectasis, pulmonary thromboembolism, etc.) or other severe systemic disease（myocardial infarction, malignant tumor, etc.）
* had a poor cooperation to the test or limited understandings, were immunocompromised, or had participated other clinical trials for the past 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
whether there was improvement in weekly PEFR | from commencement of LTRA therapy to (28±7) days
  The primary outcome was a qualitative measure, with the results being expressed as either yes or no ('1' or '0' in Logistic model).PEFR was defined as the changed rate of peak expiratory flow, which was calculated using the formula according to maximal PEF (PEFmax) and minimal PEF (PEFmin) measured by portable PEF monitor: 100%*(PEFmax-PEFmin)/[(PEFmax+PEFmin)*1/2]. A higher PEFR is more suggestive of instability of asthma control.

SECONDARY OUTCOMES:
whether there was improvement in post- treatment FENO | from commencement of LTRA therapy to (28±7) days
  In Logistic regression model, whether there was improvement shown in post-treatment FENO as compared with pre-treatment level was expressed as either 'yes' or 'no', with symbols of '1' or '0'. Thus the measure was qualitative one. FENO represented fractional exhaled nitric oxide above.
whether there was improvement in post- treatment PEF max | from commencement of LTRA therapy to (28±7) days
  In Logistic regression model, whether there was improvement shown in post-treatment PEFmax as compared with pre-treatment level was expressed as either 'yes' or 'no', with symbols of '1' or '0'. Thus the measure was qualitative.
whether there was improvement in post- treatment PEF min | from commencement of LTRA therapy to (28±7) days
  In Logistic regression model, whether there was improvement shown in post-treatment PEFmin as compared with pre-treatment level was expressed as either 'yes' or 'no', with symbols of '1' or '0'. Thus the measure above was qualitative.
whether there was improvement in post- treatment PD20FEV1-LTD4 | from commencement of LTRA therapy to (28±7) days
  In Logistic regression model, whether there was improvement shown in post-treatment PD20FEV1-LTD4 as compared with pre-treatment level was expressed as either 'yes' or 'no', with symbols of '1' or '0'. Thus the measure above was qualitative. PD20FEV1-LTD4 referred to as the provocative dosage causing a 20% fall in FEV1 while using Leukotriene D4 as a bronchoprovocant.
whether there was improvement in post- treatment PD20FEV1-MCh | from commencement of LTRA therapy to (28±7) days
  In Logistic regression model, whether there was improvement shown in post-treatment PD20FEV1-MCh as compared with pre-treatment level was expressed as either 'yes' or 'no', with symbols of '1' or '0'. Thus the measure above was qualitative. PD20FEV1-MCh referred to as the provocative dosage causing a 20% fall in FEV1 while using methacholine as a bronchoprovocant.
whether there was improvement in post- treatment AQLQ symptom score | from commencement of LTRA therapy to (28±7) days
  In Logistic regression model, whether there was improvement shown in post-treatment AQLQ symptom score as compared with pre-treatment level was expressed as either 'yes' or 'no', with symbols of '1' or '0'. Thus the measure above was qualitative. Items with regard to asthma symptoms were extracted from the whole AQLQ score, with the total score of 84. Higher score represented better asthma control.
whether there was improvement in post- treatment ACT score | from commencement of LTRA therapy to (28±7) days
  In Logistic regression model, whether there was improvement shown in post-treatment ACT score as compared with pre-treatment level was expressed as either 'yes' or 'no', with symbols of '1' or '0'. Thus the measure above was qualitative. The total score of ACT was 25, with 5 questions in all. Higher score was indicative of better asthma control.
whether there was improvement in pre-challenge FEV1 | from commencement of LTRA therapy to (28±7) days
  In Logistic regression model, whether there was improvement shown in post-treatment pre-challenge FEV1 as compared with pre-treatment level was expressed as either 'yes' or 'no', with symbols of '1' or '0'. Thus the measure was qualitative one.
whether there was a gradual decrease in weekly use of salbutamol | from commencement of LTRA therapy to (28±7) days
  In Logistic regression model, whether there was a gradual decrease in weekly use of salbutamol as compared with pre-treatment level was expressed as either 'yes' or 'no', with symbols of '1' or '0'. Thus the measure was qualitative one.
the days without using salbutamol | from commencement of LTRA therapy to (28±7) days
  This was a quantitative parameter
monthly PEFR | from commencement of LTRA therapy to (28±7) days
  This was a quantitative parameter, which was expressed as percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Guan WJ, Shi X, Zheng JP, Gao Y, Jiang CY, Xie YQ, Liu QX, Zhu Z, Guo E, An JY, Yu XX, Liu WT, Zhong NS. Leukotriene D4 inhalation challenge for predicting short-term efficacy of montelukast: a pilot study. Clin Respir J. 2015 Jan;9(1):111-20. doi: 10.1111/crj.12117. Epub 2014 Mar 5. PMID 24506412